CLINICAL TRIAL: NCT00681759
Title: A Prospective Descriptive, Multi-National, Multi-Centre Observational Study of Burden of Upper GI-Symptoms in Subjects With Cardiovascular Risk or Disease Receiving Treatment With Low-Dose Aspirin
Brief Title: An Observational Study of Burden of Upper GI-Symptoms in CV Risk Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD, Medical Science Director, Nexium, AstraZeneca Pharmaceuticals
Other Study IDs: D961FC00004
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Cardiovascular Disease
Keywords: Low Dose Aspirin (LDA); Cardiovascular disease; Low Dose Aspirin (LDA) use in in subjects with cardiovascular risk or disease
MeSH Terms: conditions — Cardiovascular Diseases; Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients who have been prescribed Low Dose Aspirin (LDA) usage in the past 12 months, or those about to begin LDA, will complete a one-time in-office survey using an electronic personal digital assistant (PDA) device (termed SitePro).
- 2: 420 subjects stratified into three groups varying on length of time using Low Dose Aspirin (LDA)
- 3: Up to 20 subjects from the three EMA groups will be interviewed to further debrief their experience with Low Dose Aspirin (LDA) and upper GI symptoms.

SUMMARY:
The purpose of this study is to investigate the burden of upper gastrointestinal symptoms in patients with cardiovascular disease taking low dose aspirin

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written inform consent.
* Physician prescribed or recommended daily intake of Low Dose Aspirin (LDA) (75-325 mg daily) for cardiovascular disease prevention within the past 12 months.
* Established cardiovascular disease, such as CAD (CoronaryArtery Disease), previous TIA (Transient Ischemic Attack), ischemic stroke or subjects with known risk factors for cardiovascular disease without having experienced cardiovascular events

Exclusion Criteria:

* Need for concomitant treatment with a non-ASA NSAID (Nonsteroidal Antiinflammatory Drugs) including acyclooxygenase-2 (COX-2) selective NSAID. Occasional use of up to 1 day/week is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiovascular risk or disease receiving LDA treatment in specialist and primary care clinics.
Sampling Method: Probability Sample
Enrollment: 1836 (Actual)
Dates: Start 2008-01; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Cross-sectional survey, SitePro Survey Domains including; background, UGI screening, PPI and H2 blocker usage, interaction between UGI and LDA ,UGI symptoms, HADS, Morisky Medication Taking Behavior Scale, SF12, SSA-P | Once at enrollment

SECONDARY OUTCOMES:
EMA assessments including: Sleep, Mood, Activities, Eating/food,GI symptoms,GI coping strategies, Medication usage, Healthcare Utilization | Four times daily for three months

CONTACTS AND LOCATIONS:
Locations (3):
- Research Site, Brentwood, Tennessee, United States
- Research Site, Saint-Laurent, Quebec, Canada
- Research Site, Paris, France

REFERENCES:
- [Derived] Bytzer P, Pratt S, Elkin E, Naesdal J, Sorstadius E. Burden of upper gastrointestinal symptoms in patients receiving low-dose acetylsalicylic acid for cardiovascular risk management: a prospective observational study. Am J Cardiovasc Drugs. 2013 Feb;13(1):27-35. doi: 10.1007/s40256-012-0001-4. PMID 23315343
- [Derived] Pratt S, Thompson VJ, Elkin EP, Naesdal J, Sorstadius E. The impact of upper gastrointestinal symptoms on nonadherence to, and discontinuation of, low-dose acetylsalicylic acid in patients with cardiovascular risk. Am J Cardiovasc Drugs. 2010;10(5):281-8. doi: 10.2165/11584410-000000000-00000. PMID 20666569